CLINICAL TRIAL: NCT00504114
Title: MR Imaging of Knee Osteoarthritis and Acute Knee Injuries
Status: Completed | Type: Observational
Sponsor: University of California, San Francisco (Other)
Collaborators: National Institutes of Health (NIH) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2R01AR046905 (NIH)
Record Dates: First submitted 2007-07-17; First posted 2007-07-19 (Estimated); Last update posted 2013-12-12 (Estimated); Status verified 2013-12

CONDITIONS: Osteoarthritis, Knee
Keywords: Osteoarthritis, knee; anterior cruciate ligament; Magnetic Resonance Imaging
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Bone/cartilage tissue will be collected after the total knee replacement surgery. The tissue will further studied using advanced MR imaging techniques.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- 1: Healthy volunteers without knee pain.
- 2: Patients with mild arthritic symptoms and radiographic changes (Kellgren Lawrence score of 1, 2)
- 3: Patients with severe pain and functional limitations associated with knee arthritis (Kellgren Lawrence score of 3, 4).
  Interventions: Procedure: Total Knee Replacement
- 4: Patients with acute anterior cruciate ligament (ACL) injuries with associated osseous contusion.
  Interventions: Procedure: ACL Reconstruction Surgery
- 5: Patients with posttraumatic knee injury or degenerative condition and will have cartilage resurfacing procedures.
  Interventions: Procedure: Cartilage Resurfacing Surgery

INTERVENTIONS:
Procedure: ACL Reconstruction Surgery
  Groups: 4
Procedure: Cartilage Resurfacing Surgery
  Groups: 5
Procedure: Total Knee Replacement
  Groups: 3

SUMMARY:
The purpose of this study is to use better magnetic resonance imaging (MRI) techniques to examine the knee and the bony and soft tissue changes so as to better predict the progression of osteoarthritis and acute knee injuries.

DETAILED DESCRIPTION:
The study will examine the pathophysiology of bone marrow changes, relationship between trabecular bone and cartilage changes; and evaluate T1p relaxation methods and its' relating to cartilage loss. The protocol is geared towards sequences utilizing 3 Tesla magnetic resonance imaging (MRI) that will enable the measures of cartilage volume and T2. Measures cartilage volume and T2 are more established MR methods for studying osteoarthritis (OA).

All OA and Anterior cruciate ligament (ACL) subjects will undergo MR imaging of the knee joint at 3 Tesla at baseline,, and three annual follow up time points. Regions of interest will include the total tibial and femoral cartilage, and sub-division such as the medial and lateral compartments of the tibial and femoral cartilage to account for localized disease activity and progression.

Bone marrow edema size, MR spectroscopy based marrow fat/water content, and trabecular bone microarchitecture underlying the edema will be measured in the OA and ACL groups to determine whether there is any distinction between these measures in OA and in traumatic ACL injury, cross-sectionally and longitudinally, and their relation to cartilage loss and OA progression.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers will have had no previous knee symptoms or surgery
* Patients with mild arthritic symptoms and Kellgren Lawrence score of 2
* Patients with severe arthritic symptoms and Kellgren Lawrence score of 3, or 4
* Patients with acute ACL injury with associated bone contusion and bone edema
* Patients with posttraumatic knee injury or degenerative condition and will have cartilage resurfacing procedures
* Patient is willing to participate in the proposed study as evidenced by providing written informed consent.

Exclusion Criteria:

* Current use of an investigational drug
* Conditions other than OA which limit lower extremity function and mobility and/or would confound the evaluation of function (e.g., clinically significant spinal disc degeneration, painful or dysfunctional feet, peripheral vascular disease, lumbar radiculopathy or a stroke.)
* Patients with metallic fragments in the eyes, vascular clips, pacemakers, and other contraindications to MRI

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Recruitment flyers are posted at different UCSF campuses and those staff and students. Patient eligibility will determined initially bye the referring orthopedist.
Sampling Method: Non-Probability Sample
Enrollment: 139 (Actual)
Dates: Start 2006-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Pathophysiology of bone marrow changes, relationship between trabecular bone and cartilage changes | Baseline, 1 year, 2 year, 3 year

SECONDARY OUTCOMES:
Evaluate T1rho relaxation methods and its' relation to cartilage loss | Baseline, 1 year, 2 year, 3 year

CONTACTS AND LOCATIONS:
Overall Officials: Sharmila Majumdar, Ph.D., Principal Investigator — University of California, San Francisco
Locations (1):
- University of California, San Francisco; MR Surbeck Laboratory of Advanced Imaging, San Francisco, California, United States